CLINICAL TRIAL: NCT05555849
Title: Reverse Cardiac Remodeling Among Elite Athletes After Short and Long-term Detraining
Acronym: Remod
Status: Completed | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Hanne Kruuse Rasmusen, Associate professor, Bispebjerg Hospital
Other Study IDs: H-21043707
Record Dates: First submitted 2022-07-19; First posted 2022-09-27 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-03

CONDITIONS: Athlete Heart; Arrhythmias, Cardiac
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study group, Newly retired elite athletes: Elite athletes at the time of retirement of professional career. Reinvestigated after three months and thereafter yearly.

SUMMARY:
Exercise has many well-documented effects in the prevention or treatment of disease, but recently some studies have raised awareness of the possible negative effects of too much exercise. In former elite endurance athletes, an increased risk of cardiac fibrosis and arrhythmias have been described. Whether exercise itself is the culprit remains to be explored.

The right cardiac ventricle can be overloaded during long-term intense exercise, due to increased volume load and possibly an increased afterload. In a subgroub of athletes the appearance with morphological and functional changes resembling an ARVC like phenotype. Furthermore, atrial fibrillation among male middle-aged athletes is up to 5 times more common compared to age-matched non-athletes. The working hypothesis of this study is that male athletes remodel more than females and that some of thise changes are already measureable early after end of elite sporting carreer.

In this prospective cohort study, of 50 elite athletes at retirement, after 3 months and thereafter yearly for five years, to determine the characteristics of remodeling of the heart focusing on the left atrial and right ventricle.

DETAILED DESCRIPTION:
A prospective cohort study of reverse cardiac remodeling in recently retired elite athletes

Aim To explore the remodeling of the heart focusing on right ventricle and left atria as well as pulmonary circulation in elite athletes at rest and during exercise as well as the effect of short and long-term reverse remodeling after the end of a professional sporting career

Methods The investigators will initiate a 5-year longitudinal study of cardiac detraining in 50 former elite athletes.

Primary outcome Change in left atrial minimum size after three months retirement (mL)

Secondary outcome:

* Change in left atrium (LA) function measured by strain and volume measures by echocardiography and magnetic resonance cor (MRc) after three months and the following years
* Change in right and left ventricle size and function by echocardiography and magnetic resonance cor (MRc) after three months and the following years
* Change in VO2max after three months and the following years
* Change in diurnal ventricular and supraventricular ectopy and heart rate variability after three months and the following years
* Change in blood pressure, BMI after three months and the following years
* Change in plasma lipids and HbA1c after three months and the following years

The full list of examinations includes:

* Baseline family history, medical and training history
* Cardio-pulmonary exercise test
* 24-hour Holter monitoring
* Biochemistry
* Cardiac MR including contrast at rest and during exercise
* Trans thoracic echocardiography

Project organization and partners Recruitment of participants is organized in cooperation with the danish national elite sports organization (Team Danmark), Divisionsforeningen (The association of professional football clubs), and Spillerforeningen (The union of professional football players).

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years at the time of screening
* Former elite athlete from endurance sport discipline
* End of elite sporting career >1 year ago

Exclusion Criteria:

* Any known cardiac disease
* Any condition (eg, psychiatric illness) or situation that, in the investigator's opinion, could impose the subject at significant risk, or interfere significantly with the subject's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self representation of gender identity
Study Population: Healthy danish elite athletes over the age of 18, who recently retired from elitesports.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Left atrial minimum volume | 5 years
  Primary endpoint The primary aim is to assess the long-term effect on remodeling of left atrium size measured by 2D echocardiography
  • Primary endpoint: Change in LA minimum volume (mL)

CONTACTS AND LOCATIONS:
Overall Officials: Hanne K Rasmusen, ph.d., Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg-Frederiksberg Hospital, Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
Registration After the provision of informed consent, each subject will be registered in a logged web-based register (REDCap). A list of registered participants will be kept linking the subject identification number. This list will be entered in a separate database and data will be encrypted. Information will not be passed on to a third party. Bispebjerg-Frederiksberg department of cardiology supervised by consultant doctor Hanne Kruuse Rasmusen will have the overall ownership and intellectual property rights to data collected in during this project.

REFERENCES:
- [Derived] Aaroee M, Tischer SG, Christensen R, Sajadieh A, Dall CH, Thune JJ, Rasmusen H. Long-term left atrial adaptations to reduced training load in former elite athletes: a long-term follow-up longitudinal observational study. BMJ Open Sport Exerc Med. 2025 Apr 3;11(2):e002379. doi: 10.1136/bmjsem-2024-002379. eCollection 2025. PMID 40191843